CLINICAL TRIAL: NCT05305235
Title: Development of a Digital Therapeutic Targeting Anxiety Sensitivity to Reduce Posttraumatic Stress in Women Presenting for Emergency Care After Sexual Assault
Brief Title: RCT for Innovating Stress-related eHealth
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-3494
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Posttraumatic Stress Disorder; Sexual Assault; Pain
Keywords: Clinical Trials, Randomized; Prevention; eHealth; Anxiety Sensitivity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Pain

STUDY DESIGN:
Intervention Model Description: Randomization tables will be generated by the study Biostatistician and uploaded into the study REDCap database by a UNC Research Coordinator prior to launching data collection. Participants are randomized (1:1) to receive either the RISE Guide (experimental) condition or Breathe2Relax (control) condition after completing their 1-week survey. The list of assignments will be stored securely in REDCap.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be masked to their study conditions, as branding is visible in both RISE Guide and Breathe2Relax. Moreover, the UNC Research Coordinators will not be masked to condition, as they will be responsible for tracking RISE Guide progress and managing participant payments. The Principal Investigator, Biostatistician, Site Principal Investigators, Site Research Associates, and anyone involved in data analysis will remain masked to condition until data analysis is complete; masking will be maintained through reduced data viewing privileges in REDCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- RISE Guide (Experimental): The RISE (RCT for Innovating Stress-related eHealth) Guide is based on Cognitive Anxiety Sensitivity Treatment (CAST), an anxiety sensitivity intervention effective in reducing anxiety sensitivity, posttraumatic stress, depression, and anxiety. RISE Guide delivers psychoeducation and cognitive-behavioral therapy principles in an interactive, audio-visual format discussing the stress response, myth-busting cognitive distortions related to stress, and facilitating safe exposure to feared sensations. Participants then complete a validated cognitive bias modification (CBM-I) for interpretation biases related to anxiety sensitivity. Finally, intervention principles are reinforced using ecological momentary intervention (EMI), in which surveys and personalized reminders are delivered based on symptoms reported during ecological momentary assessments (EMAs)
  RISE Guide delivered by smartphone via Qualtrics and is completed in ~45 minutes over 2 weeks, with EMI weeks 1-7 post-assault.
  Interventions: Device: RISE Guide
- Relaxation Control (Active Comparator): Breathe2Relax is a mobile application that instructs users on diaphragmatic breathing, a coping tool in which slow breathing through the diaphragm reduces anxiety. Participants in the control condition will download Breathe2Relax to their smartphones and receive short message service (SMS) reminders to engage with the app. The control intervention is expected to reduce symptoms, but not as much as the cognitive-behavioral therapy strategies taught in RISE Guide.
  Interventions: Device: Relaxation Control

INTERVENTIONS:
Device: RISE Guide — Smartphone-based intervention that uses Cognitive Bias Modification to change perceptions of stress.
  Other Names: RCT for Innovating Stress-related eHealth
  Arms: RISE Guide
Device: Relaxation Control — Guides users through relaxation techniques.
  Other Names: Breathe2Relax
  Arms: Relaxation Control

SUMMARY:
The Randomized Control Trial for Innovating Stress-related eHealth (RISE) Study tests the hypotheses that a highly promising digital therapeutic (RISE Guide) targeting anxiety sensitivity (AS) will be acceptable to women sexual assault survivors; reduce survivors' anxiety sensitivity, and, in turn, posttraumatic stress.

If successful, RISE Guide could be provided at no cost to all women who present to US emergency departments for emergency care after sexual assault.

DETAILED DESCRIPTION:
The RISE Study plans to recruit up to 60 women (natal and self-identifying) who present for Sexual Assault Nurse Examiner (SANE) care within 72 hours of experiencing sexual assault. Willing participants will complete enrollment procedures (i.e., consent forms and initial survey) during this same, initial SANE care visit.

All enrolled participants will complete 4/day ecological momentary assessments (EMAs; day 1 through day 49) and complete a follow-up assessment at week 1. More information on EMA and week 1 assessment content is available in the "Outcome Measurements" section of this listing.

Following their week 1 survey, all participants will be randomized into either the active (RISE Guide) or control (Breathe2Relax app) condition. Participants will receive a link to their assigned intervention. Participants in the active condition will additionally begin receiving ecological momentary interventions (EMIs) at the end of their ecological momentary assessments, which consist of personalized feedback based on symptoms reported during EMAs.

All participants will receive an Empatica wristband in the mail. Participants will wear the wristband week 1 through week 7 and press a button on the wristband's interface whenever they experience internal (e.g. thought) or external (e.g. seeing the assailant in public) trauma reminders. The wristband will collect continuous data on participants' heart rate, temperature, and perspiration, which will be used as measurements of stress reactivity.

All participants will complete further follow-up assessments at week 7, month 6, and month 12.* More information on each follow-up assessment's content is available in the "Outcome Measurements" section of this listing.

*The month 12 follow-up assessment was removed via an IRB modification approved on December 14, 2022. Participants enrolled after December 14, 2022 will not complete this timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Women sexual assault survivors presenting for emergency care <72 hours post-assault at one of our study locations.
* English speakers
* 18+ years of age
* Able to provide informed consent
* Have a smartphone with continuous service >1 year

Exclusion Criteria:

* Inability to provide informed consent (e.g., serious injury preventing the ability to hear, speak, or see to consent and participate, or other causes (e.g., diagnosed cognitive deficits, diagnosed dementia, asleep at time of screening).
* Prisoner
* Currently pregnant
* Lives with assailant and plans to continue to do so
* Admitted patient
* No mailing address
* Previously enrolled
* No SANE examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as woman.
Enrollment: 75 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A. McLean, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Nicole A. Short, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, SANE Program, Chapel Hill, North Carolina
  - Austin Stop Abuse for Everyone (SAFE), Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared by reasonable request beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available 9 to 36 months following publication and will remain available for five years.
Access Criteria: The investigator who proposes to use the data has IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Broderick JE, DeWitt EM, Rothrock N, Crane PK, Forrest CB. Advances in Patient-Reported Outcomes: The NIH PROMIS((R)) Measures. EGEMS (Wash DC). 2013 Aug 2;1(1):1015. doi: 10.13063/2327-9214.1015. eCollection 2013. PMID 25848562
- [Derived] Short NA, Pezza M, Reyes LD, Black J, Serrano K, McLean SA. The role of posttraumatic stress disorder symptoms in pain severity, interference, and variability after sexual assault: An ecological momentary assessment study. J Psychopathol Clin Sci. 2025 Dec 11:10.1037/abn0001083. doi: 10.1037/abn0001083. Online ahead of print. PMID 41379700

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 75 participants who signed informed consent, only 60 completed the required one-week follow up and were randomly assigned to a treatment intervention.
Groups:
- RISE Guide: The RISE (RCT for Innovating Stress-related eHealth) Guide is based on Cognitive Anxiety Sensitivity Treatment (CAST), an anxiety sensitivity intervention effective in reducing anxiety sensitivity, posttraumatic stress, depression, and anxiety. RISE Guide delivers psychoeducation and cognitive-behavioral therapy principles in an interactive, audio-visual format discussing the stress response, myth-busting cognitive distortions related to stress, and facilitating safe exposure to feared sensations. Participants then complete a validated cognitive bias modification (CBM-I) for interpretation biases related to anxiety sensitivity. Finally, intervention principles are reinforced using ecological momentary intervention (EMI), in which surveys and personalized reminders are delivered based on symptoms reported during ecological momentary assessments (EMAs)
  RISE Guide delivered by smartphone via Qualtrics and is completed in ~45 minutes over 2 weeks, with EMI weeks 1-7 post-assault.
  RISE Guide: Smartphone-based intervention that uses Cognitive Bias Modification to change perceptions of stress.
Period: Overall Study
Arm/Group | RISE Guide | Relaxation Control
Started | 27 | 33
Completed | 19 | 17
Not Completed | 8 | 16

BASELINE CHARACTERISTICS:
Groups:
- RISE Guide: The RISE (RCT for Innovating Stress-related eHealth) Guide is based on CAST, an anxiety sensitivity intervention effective in reducing anxiety sensitivity, posttraumatic stress, depression, and anxiety. RISE Guide delivers psychoeducation and cognitive-behavioral therapy principles in an interactive, audio-visual format discussing the stress response, myth-busting cognitive distortions related to stress, and facilitating safe exposure to feared sensations. Participants then complete a validated cognitive bias modification (CBM-I) for interpretation biases related to anxiety sensitivity. Finally, intervention principles are reinforced using ecological momentary intervention (EMI), in which surveys and personalized reminders are delivered based on symptoms reported during ecological momentary assessments (EMAs)
  RISE Guide delivered by smartphone via Qualtrics and is completed in ~45 minutes over 2 weeks, with EMI weeks 1-7 post-assault.
  RISE Guide: Smartphone-based intervention that uses Cognitive Bias Modification to change perceptions of stress.
- Total: Total of all reporting groups
Arm/Group | RISE Guide | Relaxation Control | Total
Number analyzed (Participants) | 27 | 33 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.80 (6.90) | 25.38 (6.64) | 25.56 (6.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 17 | 22 | 39
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 17 | 21 | 38
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 33 | 60

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence/Acceptability Scale
Description: The Treatment Adherence/Acceptability Scale (TAAS) is a 10-item measure of treatment acceptability (e.g., I would recommend this treatment to a friend) and adherence (e.g., I would be able to finish [this treatment]) that participants rate on a 7-point Likert scale with scores ranging from 10-70. Higher scores indicate higher acceptability.
Time Frame: 1 Week
Population: This measure was only provided to participants in the active (RISE Guide) condition. Data are reported for all RISE Guide participants who opted to complete the TAAS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RISE Guide | Relaxation Control
Number analyzed (Participants) | 17 | 0
score on a scale | 57.53 (7.70) |

2. Secondary Outcome: Credibility/Expectancy Questionnaire
Description: Credibility/Expectancy Questionnaire (CEQ; 1 week) 6-item measure of treatment credibility and expectancy of treatment to improve symptoms. Items are rated on 9-to-11-point Likert scales. 11-point scales (0-100% in 10% intervals are recoded to align with the 1-9 scales). Higher scores indicate higher credibility/expectancy. Scores can range from 4 to 56.
Time Frame: 7 Week
Population: All data collected are reported, some were missing due to attrition. Some participants chose to opt out of certain questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RISE Guide | Relaxation Control
Number analyzed (Participants) | 21 | 22
score on a scale | 22.85 (10.98) | 18.61 (13.37)

3. Secondary Outcome: Treatment Utilization and Acceptability
Description: 6 items self-report survey created for the current study on a 5-point Likert scale, such as How often did you log in? How interested were you? and 4 open-ended questions; e.g., What did you like about RISE Guide?; What did you not like? Lower scores indicate higher treatment utilization and acceptability. Scores range from 6-30.
Time Frame: 7 Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RISE Guide | Relaxation Control
Number analyzed (Participants) | 22 | 19
score on a scale | 12.45 (4.51) | 10.89 (6.58)

4. Secondary Outcome: Average Number of Participants Successfully Randomized Per Month Over the Entirety of the Study
Description: The purpose of this outcome is to measure feasibility across the entirety of successful recruitment and randomization.
Time Frame: From first to last participant approached (up to 20 months)
Measure: Mean (Standard Deviation); unit: Participants recruited and randomized
Groups:
- All Participants Enrolled and Randomized: Participants who were enrolled and randomized regardless of treatment condition.
Arm/Group | All Participants Enrolled and Randomized
Number analyzed (Participants) | 60
Participants recruited and randomized | 2 (2.52)

5. Secondary Outcome: Final Proportion of Participants Who Completed Follow-ups
Description: The proportion of participants who complete follow-ups (i.e., 7-week, 6 months) will be used to evaluate feasibility of retaining the target sample (goal retention=75% or higher).
Time Frame: 7 Weeks Follow Up, 6 Month Follow Up (up to 7 months)
Measure: Number; unit: proportion of participants
Arm/Group | RISE Guide | Relaxation Control
Number analyzed (Participants) | 27 | 33
proportion of participants
  7 Weeks | 0.85 | 0.67
  6 Months | 0.70 | 0.52

6. Secondary Outcome: Unexpected Adverse Events by Event
Description: Investigators will examine whether unexpected adverse events occur throughout each participant's participation in the study.
Time Frame: up to approximately 7 months
Measure: Number; unit: adverse events
Arm/Group | RISE Guide | Relaxation Control
Number analyzed (Participants) | 27 | 33
adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 6-month follow-up, up to 7 months total.
Arm/Group | RISE Guide | Relaxation Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/33
Other Adverse Events (participants affected / at risk) | 0/27 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT05305235/Prot_SAP_000.pdf